CLINICAL TRIAL: NCT02546531
Title: Phase I Study of Defactinib Combined With Pembrolizumab and Gemcitabine in Patients With Advanced Cancer
Brief Title: Defactinib Combined With Pembrolizumab and Gemcitabine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); Merck Sharp & Dohme LLC (Industry); Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201510157
Record Dates: First submitted 2015-08-14; First posted 2015-09-11 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Advanced Solid Tumors; Solid Tumors; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — defactinib; pembrolizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (defactinib, pembrolizumab, gemcitabine) (Experimental): * Defactinib is an oral drug which will be administered on an outpatient basis at the prescribed dose twice a day daily during each 21-day cycle.
  * Pembrolizumab is an intravenous (IV) drug which will be administered on an outpatient basis over 30 minutes (-5/+10) at a dose of 200 mg on Day 1 of each 21-day cycle.
  * Gemcitabine is an IV drug which will be administered on an outpatient basis over 30 minutes at the prescribed dose on Days 1 and 8 of each 21-day cycle.
  * Participants enrolled in Dose Level 1 and 2 will not receive gemcitabine.
  Interventions: Biological: Defactinib; Biological: Pembrolizumab; Drug: Gemcitabine
- Dose expansion (defactinib, pembrolizumab, gemcitabine) (Experimental): * Defactinib is an oral drug which will be administered on an outpatient basis at the prescribed dose twice a day daily during each 21-day cycle.
  * Pembrolizumab is an intravenous (IV) drug which will be administered on an outpatient basis over 30 minutes (-5/+10) at a dose of 200 mg on Day 1 of each 21-day cycle.
  * Gemcitabine is an IV drug which will be administered on an outpatient basis over 30 minutes at the prescribed dose on Days 1 and 8 of each 21-day cycle.
  * Participants enrolled in Dose Level 1 and 2 will not receive gemcitabine.
  Interventions: Biological: Defactinib; Biological: Pembrolizumab; Drug: Gemcitabine

INTERVENTIONS:
Biological: Defactinib
  Other Names: VS-6063
Biological: Pembrolizumab
  Other Names: Keytruda; MK-3475
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
In pancreatic cancer, targeting the tumor microenvironment has become a promising therapeutic strategy. Focal adhesion kinase (FAK) pathway activation is essential for promoting a fibrotic and inflammatory tumor microenvironment, and FAK inhibitors have demonstrated reasonable anti-tumor activity in the preclinical setting. Furthermore, a maximal synergetic effect was achieved when a FAK inhibitor was given in combination with a PD-1 antagonist and chemotherapy in multiple pancreas tumor animal models. This supports the concept of using FAK inhibitors to reduce stromal fibrosis during checkpoint immunotherapeutic treatment. Therefore, these robust preclinical findings will be tested in the proposed phase I trial.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation cohort: Histologically or cytologically confirmed diagnosis of advanced solid tumor for which standard curative or palliative measures do not exist or are no longer effective.
* Expansion cohort: Histologically or cytologically confirmed diagnosis of advanced pancreatic cancer.

  * Maintenance group (n=10): Patients must be stable on front-line therapy (defined as at least 4 months stable disease on nab-paclitaxel + gemcitabine)
  * Second-line group (n=10): Patients must have failed or could not tolerate the front line of 5FU-based therapy for advanced pancreatic cancer at least one line of chemotherapy indicated for advanced pancreatic cancer
* Expansion cohort: There should be a 2 to 4 week break between the patient's last dose of standard chemotherapy to initiation of the first cycle of study drugs. Longer than 4-week break may be permitted at the discretion of the PI.
* Expansion cohort: No more than one line of prior systemic therapy for advanced pancreatic adenocarcinoma allowed
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Life expectancy > 3 months
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN, or ≤ 5.0 x IULN if due to liver involvement by tumor
  * Creatinine ≤ 1.5 x IULN or glomerular filtration rate of ≥ 60 mL/min
  * INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
* Corrected QT interval (QTc) < 480 ms (as calculated by the Fridericia correction formula).
* Women of childbearing potential and men must agree to use adequate contraceptive methods prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy ≤ 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* No clinically evident ascites that requires therapeutic paracentesis.
* At risk of bowel perforation
* Prior treatment with a drug of the FAK inhibitor class or with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior treatment with systemic gemcitabine less than 6 months
* Currently receiving any other investigational agents
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to defactinib, pembrolizumab, gemcitabine, or other agents used in the study.
* Received a live vaccine within 30 days prior to the first study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
* Has an active autoimmune disease requiring systemic treatment within the past 2 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidisms stable on hormone replacement or Sjorgen's syndrome would not e excluded from the study.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Major surgery within 28 days prior to the first study treatment.
* History or evidence of cardiac risk including any of the following: history or evidence of current clinically significant uncontrolled arrhythmias or arrhythmia requiring treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia; history of acute coronary syndromes within 6 months prior to the first dose of study therapy (including myocardial infarction and unstable angina, coronary angioplasty, or stenting); or any history of congestive heart failure with most recent ejection fraction < 45% (screening LVEF assessment without history of CHF is not required).
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected)
* Requires continued use of warfarin for anticoagulation and cannot stop warfarin or be safely switched to another anticoagulant
* Gastrointestinal condition that could interfere with the swallowing or absorption of study medication.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, immunosuppression, autoimmune conditions, underlying pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pembrolizumab and/or defactinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose | Completion of the first cycle of all patients enrolled (approximately 25 months)
  * The recommended phase II dose will be determined from the maximum tolerated dose (MTD) found in the dose escalation cohort.
  * The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle (21 days). Dose escalations will proceed until the MTD has been reached or the completion of cycle 5.

SECONDARY OUTCOMES:
Safety and toxicity as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 30 days after completion of treatment (estimated average of 7 months)
Objective response rate (ORR) in dose escalation cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  * The definition of ORR is the proportion of patients who achieved a complete response or a partial response
  * The definition of complete response (CR) is the disappearance of all target lesions, non-target lesions, and no new lesions
  * The definition of partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions and no new lesions
Objective response rate (ORR) in dose expansion cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  * The definition of ORR is the proportion of patients who achieved a complete response or a partial response
  * The definition of complete response (CR) is the disappearance of all target lesions, non-target lesions, and no new lesions
  * The definition of partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions and no new lesions
Treatment duration in dose escalation cohort | Completion of treatment (estimated average of 6 months)
Treatment duration in dose expansion cohort | Completion of treatment (estimated average of 6 months)
Progression-free survival (PFS) in dose escalation cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one more new lesions
Progression-free survival in dose expansion cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one more new lesions
Overall survival (OS) in dose escalation cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  -OS: duration of time from start of treatment to time of death from any cause
Overall survival in dose expansion cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
  -OS: duration of time from start of treatment to time of death from any cause
Immune-related PFS in dose escalation cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)
Immune-related PFS in dose expansion cohort | Up to 2 years after completion of treatment (estimated average to be 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu